CLINICAL TRIAL: NCT04239079
Title: Autoimmune Features of Neurodegenerative Disorders
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Julian P. Agin-Liebes, Assistant Professor of Neurology, Columbia University
Other Study IDs: AAAS1669; 1R01NS095 435-01A1 (Other Grant/Funding Number: National Institute of Neurological Disorders and Stroke)
Record Dates: First submitted 2020-01-21; First posted 2020-01-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Alzheimer Disease; Mild Cognitive Impairment
Keywords: Autoimmune features; Parkinson's disease; Alzheimer's disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD and Controls: 50% of the participants will be healthy controls and 50% will be patients diagnosed with Parkinson's disease
- AD/aMCI and Controls: 50% of the participants will be healthy controls and 50% will be patients diagnosed with Alzheimer's disease or Amnestic Mild Cognitive Impairment (aMCI)

SUMMARY:
This study is being conducted to better understand the role of inflammation in Parkinson's disease (PD) and Alzheimer's disease (AD). The investigators plan to recruit 30 PD, 30 AD/Amnestic Mild Cognitive Impairment (aMCI), and 60 age matched healthy controls in this study to study the role of immune response in PD and AD.

The study involves up to two study visits involving brief questionnaires and blood draw of up to 250cc (approximately 17 tablespoons) to be collected. More ways to participate, including 1) smaller amount blood donation (up to 100cc per visit for 1-2 visits); and 2) participation via tele-visit and mobile phlebotomy visits (blood donation up to 50cc, ~5 tubes, by a certified mobile phlebotomist at home/location of choice) now available.

DETAILED DESCRIPTION:
Neurodegenerative diseases are characterized by the misprocessing of specific proteins, but how and if this results in cell death is unknown. This study is being conducted to better understand the role of inflammation in Parkinson's disease (PD) and Alzheimer's disease (AD). Both AD and PD have long been known to feature prominent neuroinflammatory components. Preliminary studies have found autoimmune features in several patients including recognition of self-antigens by specific T cells. This study will test the hypothesis that AD and PD are associated with self-derived antigens (alpha-syn and tau protein) that become recognized by T cells during aging and disease. The overall aim is to identify antigenic responses associated with PD and AD. The specific aims include:

1. Identify the protein(s) or protein segments that may trigger inflammation
2. Identify the T cells (immune cells) that may recognize and kill brain cells (neurons and astrocytes)
3. Identify the genetic profile associated with this immune response (genetic analysis of the immune system)

ELIGIBILITY:
PD and age matched controls:

For PD participants (n=30):

Inclusion criteria:

* Clinical diagnosed PD based on UK Brain Bank criteria for the clinical diagnosis of PD. And must demonstrate two of the following three, as modified from BioFIND criteria: rest tremor, rigidity, or bradykinesia, with dopaminergic medication benefit
* Age at recruitment ≥ 55
* Age at motor onset > 45
* PD onset age between 50-75 years
* Willingness to have genotyping and genetic studies

Exclusion criteria:

* Atypical features indicative of a Parkinson-Plus disorder (Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Corticobasal Degeneration (CBD)) including cerebellar signs, supranuclear gaze palsy, apraxia and other cortical signs, or prominent autonomic failure, neuroleptic treatment at time of onset of parkinsonism, active treatment with a neuroleptic at time of study entry, history of repeated strokes with stepwise progression of parkinsonism, history of repeated head injury, history of definite encephalitis, prominent gait imbalance early in the course (< 5 years)
* History of Dementia
* Recent history of cancer (past 3 years), except skin cancer
* Autoimmune disease
* Disease of the immune system (e.g. chronic leukemia, HIV)
* On chronic immune-modulatory therapy (e.g. oral steroids, azathioprine, rituximab)
* Inability to provide informed consent.

For age-matched control participants (n=30):

Inclusion criteria:

* Ages ≥55 years old
* With lack of PD in first-degree blood relatives
* Montreal Cognitive Assessment (MoCA): ≥26
* Willingness to have genotyping and genetic studies

Exclusion criteria:

* Recent history of cancer (past 3 years), except skin cancer
* Autoimmune disease
* Disease of the immune system (e.g. chronic leukemia, HIV)
* On chronic immune-modulatory therapy (e.g. oral steroids, azathioprine, rituximab)
* Inability to provide informed consent

AD/aMCI and age matched controls:

For AD/aMCI participants (n=30):

Inclusion criteria:

* Clinically diagnosed mild AD/amnestic MCI. The severity will be accessed through the Clinical Dementia Rating Scale (CDR). CDR equal to 0.5 or 1 will be necessary to meet criteria. Participants with advanced AD stage will not be capable to give their consent.
* Age ≥55 years old
* Mini-Mental State Exam (MMSE): 20-26
* Willingness to have genotyping and genetic studies

Exclusion criteria:

* Other forms of dementia including frontotemporal dementia or other dementia associated with parkinsonism such as Dementia with Lewy bodies (DLB), or Parkinson's disease Dementia (PDD), Progressive Supranuclear Palsy or corticobasal degeneration.
* History of Parkinson's disease (PD)
* Recent history of cancer (past 3 years), except skin cancer
* Autoimmune disease
* Disease of the immune system (e.g. chronic leukemia, HIV)
* On chronic immune-modulatory therapy (e.g. oral steroids, azathioprine, rituximab)
* Inability to provide informed consent

For age-matched control participants (n=30):

Inclusion criteria:

* Healthy volunteers ≥55 years old
* CDR: 0
* MoCA: ≥26
* Willingness to have genotyping and genetic studies

Exclusion criteria:

* History of Parkinson's disease (PD)
* Recent history of cancer (past 3 years), except skin cancer
* Autoimmune disease
* Disease of the immune system (e.g. chronic leukemia, HIV)
* On chronic immune-modulatory therapy (e.g. oral steroids, azathioprine, rituximab)
* Inability to provide informed consent

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with clinically confirmed Parkinson's disease and age matched controls; Patients with clinically confirmed Alzheimer's disease/ amnestic Mild Cognitive Impairment and age matched controls
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with T-cell immune response | Week 1-2
  Blood samples from patients and controls will be processed. The presence of T cell response against the candidate antigens by patient blood-derived peripheral blood mononuclear cells (PBMC) will be assessed using an enzyme-linked immunosorbent spot (ELISPOT) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Marder, MD, MPH, Principal Investigator — Columbia University; David Sulzer, PhD, Principal Investigator — Columbia University; Julian P Agin-Liebes, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sulzer D, Alcalay RN, Garretti F, Cote L, Kanter E, Agin-Liebes J, Liong C, McMurtrey C, Hildebrand WH, Mao X, Dawson VL, Dawson TM, Oseroff C, Pham J, Sidney J, Dillon MB, Carpenter C, Weiskopf D, Phillips E, Mallal S, Peters B, Frazier A, Lindestam Arlehamn CS, Sette A. T cells from patients with Parkinson's disease recognize alpha-synuclein peptides. Nature. 2017 Jun 29;546(7660):656-661. doi: 10.1038/nature22815. Epub 2017 Jun 21. PMID 28636593
- [Background] Garretti F, Agalliu D, Lindestam Arlehamn CS, Sette A, Sulzer D. Autoimmunity in Parkinson's Disease: The Role of alpha-Synuclein-Specific T Cells. Front Immunol. 2019 Feb 25;10:303. doi: 10.3389/fimmu.2019.00303. eCollection 2019. PMID 30858851
- [Background] Lindestam Arlehamn CS, Garretti F, Sulzer D, Sette A. Roles for the adaptive immune system in Parkinson's and Alzheimer's diseases. Curr Opin Immunol. 2019 Aug;59:115-120. doi: 10.1016/j.coi.2019.07.004. Epub 2019 Aug 17. PMID 31430650
- [Background] Lindestam Arlehamn CS, Pham J, Alcalay RN, Frazier A, Shorr E, Carpenter C, Sidney J, Dhanwani R, Agin-Liebes J, Garretti F, Amara AW, Standaert DG, Phillips EJ, Mallal SA, Peters B, Sulzer D, Sette A. Widespread Tau-Specific CD4 T Cell Reactivity in the General Population. J Immunol. 2019 Jul 1;203(1):84-92. doi: 10.4049/jimmunol.1801506. Epub 2019 May 13. PMID 31085590
- [Background] Lindestam Arlehamn CS, Dhanwani R, Pham J, Kuan R, Frazier A, Rezende Dutra J, Phillips E, Mallal S, Roederer M, Marder KS, Amara AW, Standaert DG, Goldman JG, Litvan I, Peters B, Sulzer D, Sette A. alpha-Synuclein-specific T cell reactivity is associated with preclinical and early Parkinson's disease. Nat Commun. 2020 Apr 20;11(1):1875. doi: 10.1038/s41467-020-15626-w. PMID 32313102